CLINICAL TRIAL: NCT04930029
Title: Evaluation of Long-term Adverse Effects of Gastric Bypass in Omega
Acronym: OMEGA10
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_82; 2020-A03156-33 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2021-06-10; First posted 2021-06-18 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Bypass Complication; Obesity
Keywords: One anastomosis gastric bypass; obesity; bariatric surgery; GERD; long term
MeSH Terms: conditions — Obesity; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OAGB150: One anastomosis gastric bypass with 150cm biliary limb
  Interventions: Other: Ten year evaluation
- OAGB200: One anastomosis gastric bypass with 200cm biliary limb
  Interventions: Other: Ten year evaluation

INTERVENTIONS:
Other: Ten year evaluation — Clinical, biological and endoscopic evaluation

SUMMARY:
The omega gastric bypass (OAGB) is developing worldwide as an alternative to the Y gastric bypass (RYGB). Cases of nutrition deficiency after OAGB, in particular protein deficency, are regularly reported in the literature, raising the question of the medium/long-term safety of this procedure. In its technology assessment report issued in September 2019 (HAS, 2019), the Haute Autorité de Santé rules on the invalidity of OAGB with a 200 cm biliary limb and the lack of sufficient data on the safety of OAGB with a 150 cm biliary limb compared to RYGB. The lack of long-term data on weight, resolution of comorbidities, quality of life, and endoscopic evaluation given the risk of lower esophageal cancer is also noted.

The main objective of the study is to compare the incidence of serious adverse events related to surgery after OAGB at 10 years, according to 2 types of loop: a realization with a 150-cm biliary loop (OAGB AB150) versus a realization with a 200-cm biliary loop (OAGB AB200).

ELIGIBILITY:
Inclusion Criteria:

* Patients who received 10 ± 2 years ago (between 2009 and 2013) an OAGB with a 150 or 200cm biliary limb. Patients should be consecutive at each center.
* Patients fulfilling the criteria of indication for bariatric surgery at the time of their intervention according to the recommendations of the HAS (HAS, 2009) in an expert center.
* Patients agreeing to perform an endoscopic evaluation with biopsies at 10 years
* Patients who gave their consent
* Patients with health insurance coverage

Exclusion Criteria:

* Contraindication to bariatric surgery defined according to HAS recommendations (HAS, 2009)
* Persons deprived of liberty, under guardianship, or under curatorship
* Patients included in a protocol with a conflict of interest with OMEGA10.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study involves patients:
  * operated between 2008 and 2013 for an OAGB with a 150 or 200cm biliary limb
  * fulfilling the HAS criteria(HAS, 2009) at the time of their surgery: BMI ≥ 40 kg/m2 or BMI ≥ 35 kg/m2 associated with a comorbidity likely to be improved by weight loss
  * benefiting from a follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious surgery-related adverse events | 10 years after surgery
  A serious adverse event is defined as a medical event that requires hospitalization, is life-threatening, results in persistent or substantial disability, or results in death. The "surgery-related" character will be described by each investigator in the first instance and homogenized by the group of experts designated at the beginning of the study.

SECONDARY OUTCOMES:
incidence of serious adverse events not related to surgery | 10 years after surgery
Nutritional biological status , assessed by evaluation of malnutrition parameters | 10 years after surgery
Nutritional clinical status, assessed by dietitian evaluation | 10 years after surgery
Excess weight loss percentage | 10 years after surgery
  calculated as follows: (weight at 10 years - initial weight) / (initial weight - ideal weight) x 100 The ideal weight is defined as the weight corresponding to a BMI = 25 kg/m2. The initial weight is the weight on the day of surgery.
Metabolic comorbidities remission | 10 years after surgery
Diabetes remission | 10 years after surgery
Hypertension remission | 10 years after surgery
Obstructive sleep apnea remission | 10 years after surgery
Dyslipidemia remission | 10 years after surgery
Quality of life by BAROS score (Bariatric analysis and reporting outcome system) | 10 years after surgery
Quality of life by GIQLI score (Gastro Intestinal Quality of Life index) questionnaires | 10 years after surgery
  The GIQLI is a score to evaluate digestive disorders in 36 items, ranging from 0 (the worst quality of life) to 144 (the best quality of life).
GERD | 10 years after surgery
  GERD, assessed by clinical evaluation, PPI use, and endoscopic signs of GERD (gastritis, oesophagitis, anastomotic ulcer, Barrett's esophagus, gastric metaplasia, esophageal metaplasia

CONTACTS AND LOCATIONS:
Overall Officials: Robert CAIAZZO, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Claude Huriez - Service de chirurgie générale et endocrinienne, Lille, France